# Department of Veterans Affairs Research Information Sheet

VAAAHS Research IRB Approved 12/28/2023



Title of Study:

Enhancing Purpose and Well-Being Through a Volunteering Experience Connecting Veterans with

English Language Learners

Principal Investigator: John Piette, PhD

VAMC: VA Ann Arbor Healthcare System

You are being asked to participate in a research study conducted by John Piette at the Ann Arbor VA. We are conducting a study to address the loss of purpose, and social isolation among Veterans. The primary hypothesis is that structured contact via videocam between Veterans and English Language Learners (ELLs) using accessible technology will enhance Veterans' sense of life purpose and overall psychological well-being. Your participation in this research study is voluntary. You may choose not to participate or leave the study at any time without penalty or loss of benefits to which you were otherwise entitled.

#### WHY IS THIS STUDY BEING DONE?

We are conducting a research study to test a program called "V-SPEAK!" (Veteran Service Promoting English Acquisition and Knowledge). In this program, Veterans with symptoms of depression, anxiety, or PTSD, help English Language Learners (ELLs) improve their English skills by having conversations. The conversations take place by videoconference. As part of testing the V-SPEAK! Program, we will look at how to recruit participants, how to implement the program, how to retain participants, and the program's impact on the participants.

#### WHAT WILL HAPPEN IF I PARTICIPATE IN THIS STUDY?

If you agree to participate, you will be asked to do a baseline survey that will ask you questions about things like your general health, well-being, quality of life, loneliness, depressive symptoms, health service use, and demographic information such as your age and education level.

We are recruiting men and women who would like to help someone improve their English language skills, are at least 18 years of age or older, speak English fluently, and have internet access to connect to video conferencing software.

We plan to recruit 40 Veterans from the Ann Arbor VA and 40 English Language Learners (ELLs) from the community.

We will contact you when the next ELL is available at the times that are convenient for you. We will pair you with an English Language Learner. ELLs will be told their conversation partner has "symptoms of mood problems, such as depression or anxiety". We will use a standard videoconferencing platform such as Microsoft Teams. The first two sessions will be facilitated by study staff who will introduce each session, assist with technical issues, and ensure that both parties have their materials and are comfortable. All sessions will be video and audio recorded. Additionally, if both participants are in agreement after the second session, they can complete the following 6 sessions without a staff member monitoring their sessions. A questionnaire will be sent to you via email after each session, to allow you and your ELL partner to privately express any issues or concerns. Research staff will actively review responses after every session. They will take note of any concerns, and they will follow-up with either participant if necessary.

Before each scheduled session, you will get a reminder phone call or email. You will be asked to do a follow-up survey after your last conversation session. Your involvement in this study will last about 8 weeks. Each survey will take about 30-minutes.

Before the first conversation session, there will be a 30-minute orientation to the program with a staff member. During the orientation you will get an outline of the program, training on how to use the videoconferencing software, an outline for the conversation sessions, and tips for talking with the English Language Learner. You will get training materials and will have access to phone support from the study team for any problems during the study.

You will also be asked to complete a follow-survey with research staff over the phone or via videoconference. We will contact you to schedule and remind you about the follow-up survey. The follow-up survey will last about a half-hour and will ask you questions about topics like your well-being, quality of life, loneliness, depressive symptoms, health service use, and program satisfaction. After completing the follow-up survey, your participation in the study will be complete.

# WHAT ARE KEY REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY (BENEFITS)?

You might not receive any personal benefits from being in this study. But, if you agree to be in the study, you may get satisfaction in helping someone better their English skills. Even if you don't benefit personally, the study will help us gain information about how to make programs like this one more helpful for Veterans.

## WHAT ARE KEY REASONS YOU MIGHT CHOOSE NOT TO VOLUNTEER FOR THIS STUDY (RISKS)?

Although small, there are risks. Doing a survey or interview, or speaking with the English Language Learner, could be stressful for some people. To reduce this, you may skip any question in the survey or interview at any time, you can disconnect from any conversation session at any time, and you can contact the study team to report any stressful events or to discuss any concerns about the study. You can also withdraw from the study at any time.

There is a very small risk that people other than the study team may see your study data, or that a language learner could share information about you with someone else. There is a very small risk that data from the video conferences or the session reminders sent over phone lines or email could be intercepted by an outside party. There may be other risks that are unforeseeable at this time.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits or rights you would normally have if you choose not to volunteer.

## WHO WILL SEE MY INFORMATION AND HOW WILL IT BE PROTECTED?

The information collected for this study will be kept confidential. We will protect the confidentiality of your study records by keeping them in a restricted computer file that only authorized staff can access. This study record will not show your name but will have codes entered in it that will link the information to you. Your name and any other information that can directly identify you will be stored separately from the study data. We will keep your research record confidential, to the extent provided by federal, state, and local law.

If we write a report or article about this study or share the study data set with others, we will do so in such a way that you cannot be directly identified. No information by which you can be identified will be released or published unless required by law.

There are times when we might have to show your records to other people. For example, someone from the Office of Human Research Protections, the Government Accountability Office, the Office of the Inspector

General, the VA Office of Research Oversight, our local Research and Development Committee, and other study monitors may look at or copy portions of records that identify you.

# **Health Information Portability and Accountability Act (HIPAA)**

There are rules to protect your private information. Federal and state laws and the federal medical Privacy Rule also protect your privacy. By giving your verbal consent, you provide your permission called your 'authorization,' for the use and disclosure of information protected by the Privacy Rule.

The research team working on the study will collect information about you. This includes things learned from the procedures described in this research information sheet. The study team may also collect other information including your name, address, date of birth, and information from your medical records such as drug, alcohol use, or mental health treatment.

The research team may also need to disclose the information to others as part of the study progress. Others may include the VA Institutional Review Board, and the local VA medical facility Human Research Protections Program.

Your health information disclosed pursuant to this authorization may no longer be protected by Federal laws or regulations and may be subject to re-disclosure by the recipient. While this study is being conducted you will not have access to your research related health records. This will not affect your VA healthcare, including your doctor's ability to see your records as part of your normal care and will not affect your right to have access to the research records after the study is completed.

You can revoke this authorization, in writing, at any time. To revoke your authorization, you must write to the Principal Investigator at this facility or you can ask a member of the research team to give you a form to revoke the authorization. Your request will be valid when the Study Team receives it. If you revoke this authorization, you will not be able to continue to participate in the study. This will not affect your rights as a VHA patient to treatment or benefit outside of the study.

If you revoke this authorization, John Piette, PhD, and his research team can continue to use information about you that was collected before receipt of the revocation. The research team will not collect information about you after you revoke the authorization.

Treatment, payment or enrollment/eligibility for benefits cannot be conditioned on you signing this authorization. This authorization will expire at the end of the research study unless revoked prior to that time.

# WILL I RECEIVE ANY PAYMENT IF I PARTICIPATE IN THIS STUDY?

You will receive no payment for your participation.

# WHO CAN I TALK TO ABOUT THE STUDY?

In the event of a research related injury, the VA will provide necessary medical treatment at no cost to you unless the injury is due to noncompliance with study procedures. Please immediately contact **study staff 734-222-7671**. If you have any other questions, comments or concerns about the research, you can call or leave a voicemail message for the <u>research staff</u> at <u>734-222-7671</u>.

If you have questions about your rights as a study participant, or you want to make sure this is a valid VA study, you may contact the VA IRB Coordinator at (734) 845-3440.